CLINICAL TRIAL: NCT01966913
Title: Salvage Chemotherapy for Poor Prognosis Germ Cell Tumors - A Phase I-II Sequential Chemotherapy Protocol of Bevacizumab (Avastin) Plus High-dose ICE (Ifosfamide - Carboplatin - Etoposide) Intensification
Brief Title: Salvage Chemotherapy for Poor Prognosis Germ Cell Tumors
Acronym: TAXIFIII
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P100135
Record Dates: First submitted 2013-10-11; First posted 2013-10-22 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Germ Cell Tumor
Keywords: Germ Cell Tumors; Bevacizumab; salvage therapy
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal | interventions — Bevacizumab; ICE protocol 5

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bevacizumab (Experimental): Two intensified treatments at 6-week intervals will start on D69 (max D76) and D111 (max J118) respectively, combining:
  * A bevacizumab treatment: 7.5 mg/kg every 3 weeks from D1 to the first intensified treatment for a total of 4 injections.
  * The ICE chemotherapy regimen:
    1. Etoposide, 300 mg/m²/d in two daily injections at 12-h intervals,
    2. Carboplatin, AUC 4/d by injections adjusted daily to the creatinine clearance,
    3. Ifosfamide, 2400 mg/m²/d,
    4. For 5 consecutive days followed by HSC reinjection and G-CSF (filgrastim- Neupogen) on D11 of each intensive cycle
  Interventions: Drug: Bevacizumab; Drug: ICE chemotherapy regimen

INTERVENTIONS:
Drug: Bevacizumab
Drug: ICE chemotherapy regimen — Etoposide, 300 mg/m²/d in two daily injections at 12-h intervals, Carboplatin, AUC 4/d by injections adjusted daily to the creatinine clearance, Ifosfamide, 2400 mg/m²/d, For 5 consecutive days followed by HSC reinjection and G-CSF (filgrastim- Neupogen) on D11 of each intensive cycle

SUMMARY:
High-dose chemotherapy with autologous hematopoietic stem-cell transplantation is a standard salvage treatment used in adults with germ cell tumors (Einhorn et al, J Clin Oncol 2007).

Disease prognosis following 1 to 2 intensified combinations of etoposide - carboplatin +/- ifosfamide depends on the patient's performance status (PS) at inclusion and the prior sensitivity of the disease to cisplatin. A poor PS and/or being refractory to cisplatin suggest a higher toxicity and a bad prognosis.

However, predictive factors of response to high-dose chemotherapy do not include a chemo-sensitivity phase with a semi-intensive chemotherapy excluding a platinum compound (epirubicin - paclitaxel), which still allows stem-cell harvest. The use of this chemotherapy combination induced a response in more than one third of the patients treated during disease progression in the TAXIF I study. The same strategy was tested in the TAXIF II study, which completed the inclusion of 45 patients and was closed in May 2008. Results of the TAXIF II study, are currently being analyzed; they support the hypothesis to prioritarily treat patients with a sensitive relapsed disease at the time of the high-dose administration.

A combination of a semi-intensive sequential ICE type chemotherapy plus bevacizumab was used on a highly refractory patient. A 5 months nearly complete response was achieved. Indeed, the overexpression of VEGF (Vascular Endothelial Growth Factor) has been identified as an independent risk factor in patients with germ cell tumor. Therefore, a treatment strategy using an inductive chemotherapy followed, in case of response, by a double intensification therapy in combination with a VEGF treatment, could be an interesting approach in patients with poor prognosis germ cell tumors.

The aim of this phase I/II trial is to assess the feasibility of a Bevacizumab - ICE (Ifosfamide-Carboplatin-Etoposide) high dose combination with the support of autologous hematopoietic stem cell for two intensive consecutive cycles ("tandem" intensification) in patients with a poor prognosis germ cell tumor non refractory to a front-line mobilization chemotherapy using two half intensified consecutive combinations of Epirubicin-Paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older having signed an informed consent form.
* Germ cell tumor of gonadal origin, extra-gonadal, retro-peritoneal or primary mediastinal, excluding CNS tumors.
* Relapsed, refractory or completely refractory disease. The patients must have received:

  * For relapsed patients, two lines of a standard chemotherapy (BEP or EP in first-line treatment, VeIP or VIP in second-line treatment)
  * For refractory or completely refractory patients, one line of a standard chemotherapy (BEP or EP)
* First extra-gonadal tumor relapse
* Normal laboratory tests levels usually required for intensive treatments
* Performance status < 2.
* Life expectancy ≥ 3 months.

Exclusion Criteria:

* Brain metastases
* Lesions of growing teratoma
* Cardiovascular disease, uncontrolled hypertension
* History of transient ischemic attacks
* All other contraindications to bevacizumab treatment
* Non-healing wound, active peptic ulcer or bone fracture
* known allergy to bevacizumab or any of its excipients
* known allergy to chemotherapy including Cremophor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-04; Primary Completion 2019-03 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Response | 3 months
  Partial response or complete response evaluated by scanography and assay for tumor marker(s) a month after the end of the 2 cycles
Toxicity | 6 months
  Safety recorded according to CTCAE-v4 criteria

SECONDARY OUTCOMES:
complete response rate | within 2 years of inclusion
complete pathological response (pCR) or complete surgical response (sCR) | within 2 years after inclusion
overall survival | within 2 years after inclusion
response duration | within 2 years after inclusion
progression-free survival | within 2 years after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Tenon, Paris, France